CLINICAL TRIAL: NCT06719284
Title: Crossover Study of the Cerebral Blood Flow and Cardiac Output At Different Targeted Tidal Volumes During High Frequency Oscillation with Volume Targeted Ventilation (HFO&VTV)
Brief Title: Optimising HFO&VTV in Newborn Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 349734
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: High Frequency Oscillation; Volume Targeted Ventilation
Keywords: high frequency oscillation; volume targeted ventilation; newborn infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High frequency oscillation at the settings applied prior to the study (Active Comparator)
  Interventions: Other: HFOV at the settings applied prior to the study
- High frequency oscillation with volume targeted ventilation (Active Comparator)
  Interventions: Other: HFO&VTV at targeted tidal volumes of 1.5, 2.0 and 2.5 ml/kg in random order

INTERVENTIONS:
Other: HFO&VTV at targeted tidal volumes of 1.5, 2.0 and 2.5 ml/kg in random order — HFO&VTV at targeted tidal volumes of 1.5, 2.0 and 2.5 ml/kg in random order
  Arms: High frequency oscillation with volume targeted ventilation
Other: HFOV at the settings applied prior to the study — HFOV at the settings applied prior to the study
  Arms: High frequency oscillation at the settings applied prior to the study

SUMMARY:
Mechanical ventilation (MV) is life saving for infants requiring respiratory support in the newborn period but its use has been associated with complications. High frequency oscillation (HFO) is a type of MV that delivers small volumes of gas across the lungs at fast frequencies. HFO is a lung protective strategy but it has also been linked to brain injury due to low carbon dioxide tensions. High-frequency oscillation with volume-targeted ventilation (HFO&VTV) is a new mode of HFO in which the clinician sets a target volume of gas to be delivered to the lungs at fast rates to decrease the lung injury related to the ventilator. Further, HFO&VTV achieves better control of carbon dioxide levels and may therefore protect against brain injury. Currently, there are no written guidelines about the use of HFO&VTV. This study aim to determine the safety profile of HFO&VTV compared to HFO by comparing the velocity of blood flow to the brain in term born infants and the cardiac output in term and preterm infants during the two modes. The investigators will also determine the optimum starting value of the target tidal volume during HFOV&VTV. Infants will be studied at three different target tidal volumes for a period of 10-20 minutes each. A cranial ultrasound (for term infants only) and bedside echocardiogram will be performed at the end of each period.

DETAILED DESCRIPTION:
This is a single centre, randomised cross-over trial in newborn infants requiring high-frequency oscillatory ventilation (HFOV) at any postnatal age. Infants with known intracerebral pathology (stroke, hydrocephalus, intracerebral haemorrhage, severe HIE) and congenital cardiac abnormalities will be excluded from the study. In preterm infants cerebral blood flow will not be studied as there is no clear evidence for the significance of the resistive index (RI) in the cerebral arteries to predict brain injury and neurodevelopmental outcomes.

The research team will identify infants based on the inclusion criteria and approach parents to discuss the study and provide information leaflets.

The investigators aim to recruit a minimum of 25 infants (13 preterm and 12 term infants) over 18 months.

Informed written consent will be requested from the parents or legal guardians of the infants and the attending Neonatal Consultant will be requested to verbally assent to the study.

All infants will be oscillated using SLE6000 ventilators. Ventilation settings will be adjusted by the clinical team as per unit's protocol.

Infants will be studied when clinically stable and a blood gas confirms that the carbon dioxide (CO2) levels are in the target range (4.5 to 6.5 kPa). Participants will receive HFO&VTV at targeted tidal volumes of 1.5, 2.0 and 2.5 ml/kg in random order for a period of 10-20 minutes each. Additionally, there will be a control period of 20 minutes between each tidal volume when infants will be switched to HFOV without volume-guarantee at the settings applied prior to the study. The order in which they receive the different levels of tidal volumes will be randomised using an excel random number generator.

Transcutaneous CO2 monitoring will be applied to the infants during the study. The resistive index (RI) as an indicator of cerebral blood flow in term infants and the cardiac output of all paticipants will be assessed at the last five minutes of each twenty-minute period. Measurements of the RI and the cardiac output will also be made during the last five minutes of the control periods and the results will be averaged.

The nurse to patient ration will be according to the unit's protocol that is determined on the patient's acuity.

The investigators will also record basic epidemiologic parameters such as sex, gestational age, birth weight, mode of delivery, Apgar scores, administration of surfactant, day of life at study, mechanical ventilation starting time and HFO starting time, and initial diagnosis.

ELIGIBILITY:
Inclusion Criteria:

-Newborn infants of any gestation receiving high frequency oscillatory ventilation

Exclusion Criteria:

* Infants with known intracerebral pathology (stroke, hydrocephalus, intracerebral hemorrhage, severe hypoxic ischemic encephalopathy).
* Infants with congenital cardiac abnormalities.

Ages: 22 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The change in the Resistive Index (RI) that will be measured on term born infants using the anterior cerebral artery Doppler on cranial ultrasound | Through study completion, an average of 18 months

SECONDARY OUTCOMES:
The change in cardiac output that will be assessed with bedside ECHO in all infants | Through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Dassios, Professor, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camfferman FA, de Goederen R, Govaert P, Dudink J, van Bel F, Pellicer A, Cools F; eurUS.brain group. Diagnostic and predictive value of Doppler ultrasound for evaluation of the brain circulation in preterm infants: a systematic review. Pediatr Res. 2020 Mar;87(Suppl 1):50-58. doi: 10.1038/s41390-020-0777-x. PMID 32218536
- [Background] Tuzun F, Deliloglu B, Cengiz MM, Iscan B, Duman N, Ozkan H. Volume Guarantee High-Frequency Oscillatory Ventilation in Preterm Infants With RDS: Tidal Volume and DCO2 Levels for Optimal Ventilation Using Open-Lung Strategies. Front Pediatr. 2020 Mar 24;8:105. doi: 10.3389/fped.2020.00105. eCollection 2020. PMID 32266185
- [Background] Iscan B, Duman N, Tuzun F, Kumral A, Ozkan H. Impact of Volume Guarantee on High-Frequency Oscillatory Ventilation in Preterm Infants: A Randomized Crossover Clinical Trial. Neonatology. 2015;108(4):277-82. doi: 10.1159/000437204. Epub 2015 Sep 1. PMID 26330156
- [Derived] Kaltsogianni O, Nanjundappa M, Okoye G, Greenough A, Dassios T. Effect of different targeted tidal volumes during high-frequency oscillation with volume-targeted ventilation on cerebral blood flow velocity and cardiac output: study protocol for a randomised crossover study. Trials. 2025 Oct 22;26(1):427. doi: 10.1186/s13063-025-09179-w. PMID 41126304